CLINICAL TRIAL: NCT01016418
Title: Bovine Colostrum for Patients With Non Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Gadi Lalazar, Hadassah Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NASH Colostrum - HMO - CTIL
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Nonalcoholic Steatohepatitis; Fatty Liver Disease
Keywords: NASH; fatty liver disease; colostrum
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bovine colostrum powder (Experimental): Study treatment will consist of BCP, three 1.2 g oral tablets (equivalent to 600 mg of BCP each) for 4 weeks, from cows immunized to insulin. Patients will be followed for safety monitoring for an additional 4 weeks.
  Interventions: Dietary Supplement: Bovine colostrum powder

INTERVENTIONS:
Dietary Supplement: Bovine colostrum powder — Study treatment will consist of BCP, three 1.2 g oral tablets (equivalent to 600 mg of BCP each) for 4 weeks, from cows immunized to insulin. Patients will be followed for safety monitoring for an additional 4 weeks.

SUMMARY:
Trial Synopsis: Bovine Colostrum for patients with non alcoholic fatty liver disease (NAFLD).

Design: This is a single-arm, open-label, before-and after exploratory trial of 30 days of Bovine Colostrum Powder (BCP) to improve NAFLD and the metabolic syndrome.

Duration: 8 weeks per subject.

Sample Size: 30 subjects.

Population: Patients with biopsy proven NASH (NAS of > 4) and an ALT level of ≥ 30 (U/L).

Regimen Study treatment will consist of BCP, three 1.2 g oral tablets (equivalent to 600 mg of BCP each) for 4 weeks, from cows immunized to insulin. Patients will be followed for safety monitoring for an additional 4 weeks.

DETAILED DESCRIPTION:
1. HYPOTHESIS AND STUDY OBJECTIVES

   1.1. HYPOTHESIS

   Ingestion of bovine colostrum powder (BCP) from cows immunized to insulin will improve non alcoholic steatohepatitis and the metabolic syndrome in patients suffering from these conditions

   1.2. PRIMARY OBJECTIVES

   1.2.1 To determine the efficacy of BCP in improving liver enzyme levels in patients with NASH.

   1.2.2 To determine the safety of the administration of oral BCP to patients with NASH.

   1.3. SECONDARY OBJECTIVES

   1.3.1. To determine whether the administration of BCP will improve the metabolic syndrome in patients with NASH (namely insulin resistance).
2. INTRODUCTION

   2.1. BACKGROUND

   2.1.1. Nonalcoholic steatohepatitis.

   Nonalcoholic steatohepatitis or NASH is a common, often "silent" liver disease which affects about 2%-5% of Americans4-6. NASH is strongly associated with the metabolic syndrome, diabetes type-2 and obesity and can lead to cirrhosis, HCC, liver transplantation or death. The only mean for proving a diagnosis of NASH and separating it from simple fatty liver is liver biopsy (an invasive procedure which carries a certain degree of risk). Currently, there is no effective treatment for NASH7.

   2.1.2. The effect of Hyperimmune Bovine Colostrum on NASH

   Regulatory T cells (Tregs) are recognized as an important immunomodulatory component of the adaptive immune system. Immune dysregulation may lead to chronic inflammation, triggering chronic insulin insensitivity and non-alcoholic steatohepatitis (NASH). The role of Tregs in the adipose tissue in the regulation of NASH was not previously studied. Aim: To assess the effects of Tregs stimulation on hepatic injury and insulin resistance in NASH. Methods: Leptin deficient Ob/Ob mice were fed for 4 weeks with colostrum derived solutions (CDS) enriched with anti insulin specific antibodies (AIS-CDS, Immuron, Australia), or with purified anti insulin specific CDS (PAIS-CDS). The immunologic effect on the adipose tissue was determined by flow cytometry performed on the central adipose tissue and its stromal vasculature (SV), and compared with the effect on immune system of the liver and the spleen. Hepatic injury and insulin resistance was determined by glucose tolerance tests (GTT) and liver enzymes. Results: Oral administration of anti-insulin antibodies promoted the SV CD4+CD25+FoxP3+ cells (13.05 vs. 27.94 p=0.01). Treatment was associated with a decrease of the CD4+IL17+ lymphocyte subset in the adipose tissue (87.89 vs. 12.93, p<0.01), the SV (61.86 vs. 14.99, p<0.01), and in the liver (40.18 vs. 2.66, p<0.01). The liver CD8+CD25+FoxP3+ lymphocyte subset was significantly increased (0.36 vs. 2.39, p<0.05). The CD4/CD8+ lymphocyte ratio in the adipose tissue showed a mirror effect to that of the spleen and liver suggesting an opposite effect on lymphocyte trapping. Promotion Tregs in the adipose tissue was accompanied by a marked improvement in insulin resistance manifested by decreased glucose and insulin serum levels, and improved glucose tolerance test results (a decrease of 45%, in the area under the curve 23355 vs. 42448, in treated vs. controls, respectively), along with decreased liver enzymes (ALT levels decreased from 743.4 to 379.8 IU, p<0.05; and AST from 770.5 to 299IU, in controls vs., treated respectively, p=0.07) without a change in body weight. Conclusions: The immune system of the adipose tissue plays an important role in the regulation of the metabolic syndrome. Decreasing TH17 in the liver, adipose tissue and SV, along with promotion of CD4+CD25+FoxP3+ and CD8+CD25+FoxP3+ Tregs (in the SC and liver respectively), by oral administration of anti insulin CDS offers a new treatment modality for NASH and insulin resistance, making Tregs in adipose tissue as a new therapeutic target for alleviation of the liver damage in NASH.

   2.1.3. BCP Has Been Shown to Be Safe and Well-tolerated in Humans

   Over 80,000 packets of Anadis tabletted BCP product with the same active component has been sold in Australia over 4 years. There have been no reported adverse events reports to Anadis. BioGard itself as a higher dose separate product was approved in 2008.

   Risk of microbiological contamination: The colostrum in the product is pasteurized; strict procedures minimize risk of contamination, and tablet batches are tested for yeast, mold, coliform bacteria, Enterobacteriaceae, staphylococci, Salmonella, and Listeria. The cows for colostrum production are sourced only from bovine spongiform encephalopathy (BSE)-free countries. Additionally, milk products are considered to have no detectable infectivity and are considered unlikely to present any risk if sourced from healthy animals under the same conditions as milk collected for human consumption.

   Lactose intolerance: Bovine colostrum extract generally contains <10% lactose, compared with about 50% in normal skim milk powder; therefore, lactose intolerance is unlikely to be a major safety problem. Clinical signs can be expected in susceptible humans given 5-10g of lactose (Thorn et al, 1977). At a dose of bovine colostrum extract of 10g a day (2.8g more than the dose proposed in this study), a maximum of 1 g would be lactose.

   Side effects. No cases of death have ever been reported in studies of BCP. While the typical dose is 10g/day [8-10] doses as high as 10 g four times daily have been studied[11]. Adverse reactions have been few in number and slight in severity. In most clinical studies on the efficacy of bovine colostrum there have been no demonstrable adverse effects[9, 10, 12-15]. When they have occurred, they have mostly consisted of nausea, emesis, flatulence, and mild diarrhea[8, 11, 14, 16, 17]. In one study, transient moderate elevations in serum levels of hepatic transaminases were observed in volunteers who received bovine immunoglobulin concentrates prepared against E. coli (5/10) and rotavirus (2/10). This effect was attributed to diets high in protein provided at the hospital (13). More recently, bovine colostrum was well-tolerated in HIV-infected persons for the treatment of HIV-associated diarrhea (18).

   Colostrum administration should be avoided in person allergic to cow's milk.
3. STUDY DESIGN

   This is a single-arm, open label, before-and-after exploratory trial to evaluate the effect of 4 weeks of BCP administration on serum liver enzymes and the metabolic syndrome in patients with NASH. Candidates will be identified from among the patients treated in the department of medicine and liver unit of the Hadassah Hebrew University Medical Center and will be asked to sign an approved informed consent from before any study activities are initiated. Participants will be followed on study with weekly visits as well as for an additional 4 weeks after concluding treatment to assess safety.
4. SELECTION AND ENROLLMENT OF SUBJECTS

4.1. INCLUSION CRITERIA

4.1.1. Biopsy proven NASH (NAS score ≥ 4) 4.1.2. Serum ALT levels ≥ 30 (U/L) 4.1.3. Age 18-65 4.1.4. Treatment of diabetes by up to 2 oral medications, with stable doses for 2 months.

4.1.5. If participating in sexual activity that could lead to pregnancy, the study volunteer must agree that two reliable methods of contraception will be used simultaneously while receiving the protocol-specified medication and for 1 month after stopping the medication.

NOTE: Hormonal-based methods alone are not sufficient. At least two of the following methods MUST be used appropriately unless documentation of menopause, sterilization, or azoospermia is present:

* Condoms (male or female) with or without a spermicidal agent. - Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission
* Diaphragm or cervical cap with spermicide
* IUD
* Hormonal-based contraception

Study subjects who are not of reproductive potential (girls who have not reached menarche or women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy are eligible without requiring the use of contraceptives. Written or oral documentation communicated by clinician or clinician's staff is required by one of the following:

* Physician report/letter
* Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy)
* Discharge summary
* Laboratory report of azoospermia
* FSH measurement elevated into the menopausal range as established by the reporting laboratory.

4.1.6. Ability and willingness of subject or legal guardian/representative to provide informed consent.

1. EXCLUSION CRITERIA

i. Pregnancy or Breast-Feeding

ii. Continuous use of the following medications for more than 3 days within 30 days of study entry:

1. Immunosuppressives
2. Immune modulators
3. Systemic glucocorticoids
4. Anti-neoplastic agents
5. Insulin iii. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

iv. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.

v. Operation within the previous 3 months. vi. A serious infectious, cardiac, pulmonary, or nephrological disease vii. Allergic to cow milk or lactose intolerant.

2. STUDY TREATMENT

a. REGIMEN, ADMINISTRATION AND DURATION

i. Per-protocol treatment regimen

Subjects will receive treatment with BCP 1.8 grams (3 capsules) for 4 weeks and will then be monitored off study treatment for an additional 4 weeks.

ii. Study treatment modifications

Dose reductions will not be allowed. All study drug modifications will be documented and recorded.

b. STUDY PRODUCT FORMULATION AND PREPARATION

The study medication is supplied at tablets packaged individually in blister packs. Each 1.2 g tablet contains 600 mg of freeze-dried BCP from cows immunized to insulin as the only active component, in combination with excipients including silica colloidal anhydrous, magnesium stearate, microcrystalline cellulose and calcium carbonate. The product can be stored at room temperature and has a shelf life of 5 years.

c. PHARMACY: PRODUCT SUPPLY, DISTRIBUTION, AND ACCOUNTABILITY

i. Study product acquisition/distribution

BCP will be supplied by Immuron, and will be stored and dispensed by the research pharmacies at the Hadassah Hebrew University Medical Center.

ii. Study product accountability

The site pharmacist is required to maintain complete records of all study products.

d. CONCOMITANT MEDICATIONS

i. General guidelines

There are no specific protocol-imposed restrictions on concomitant medications, other than stipulated in the inclusion/exclusion criteria. Nonetheless, whenever a concomitant medication or study agent is initiated or a dose changed, investigators will review the concomitant medications' and study agents' most recent package inserts, investigator's brochures, or updated information from on-line sources to obtain the most current information on drug interactions, contraindications, and precautions.

ii. Prohibited medications

Use of the following medications for more than 3 days within 30 days of study entry: Insulin, immunosuppressives, immune modulators, anti-neoplastic agents, glucocorticoids.

e. ADHERENCE ASSESSMENT

At each visit, participants will be queried about the number of doses of study medication missed since the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven NASH (NAS score ≥ 4)
* Serum ALT levels ≥ 30 (U/L)
* Age 18-65
* Treatment of diabetes by up to 2 oral medications, with stable doses for 2 months
* If participating in sexual activity that could lead to pregnancy, the study volunteer must agree that two reliable methods of contraception will be used simultaneously while receiving the protocol-specified medication and for 1 month after stopping the medication.NOTE: Hormonal-based methods alone are not sufficient. At least two of the following methods MUST be used appropriately unless documentation of menopause, sterilization, or azoospermia is present:

  * Condoms (male or female) with or without a spermicidal agent. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission
  * Diaphragm or cervical cap with spermicide
  * IUD
  * Hormonal-based contraception
* Study subjects who are not of reproductive potential (girls who have not reached menarche or women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy) are eligible without requiring the use of contraceptives.
* Written or oral documentation communicated by clinician or clinician's staff is required by one of the following:

  * Physician report/letter
  * Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy)
  * Discharge summary
  * Laboratory report of azoospermia
  * FSH measurement elevated into the menopausal range as established by the reporting laboratory
* Ability and willingness of subject or legal guardian/representative to provide informed consent

Exclusion Criteria:

* Pregnancy or Breast-Feeding
* Continuous use of the following medications for more than 3 days within 30 days of study entry:

  * Immunosuppressives
  * Immune modulators
  * Systemic glucocorticoids
  * Anti-neoplastic agents
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry
* Operation within the previous 3 months
* A serious infectious, cardiac, pulmonary, or nephrological disease
* Allergic to cow milk or lactose intolerant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of BCP in improving liver enzyme levels in patients with NASH. | 4 weeks
To determine the safety of the administration of oral BCP to patients with NASH. | 8 weeks

SECONDARY OUTCOMES:
To determine whether the administration of BCP will improve the metabolic syndrome in patients with NASH (namely insulin resistance). | 4

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Unit, Hadassah, Ein Kerem, Jerusalem, Israel

REFERENCES:
- [Background] Kim JH, Jung WS, Choi NJ, Kim DO, Shin DH, Kim YJ. Health-promoting effects of bovine colostrum in Type 2 diabetic patients can reduce blood glucose, cholesterol, triglyceride and ketones. J Nutr Biochem. 2009 Apr;20(4):298-303. doi: 10.1016/j.jnutbio.2008.04.002. Epub 2008 Jul 7. PMID 18602824